CLINICAL TRIAL: NCT02446548
Title: Influence of Aliskiren on Albuminuria After Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Leszek Tylicki, Professor, Medical University of Gdansk
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ST-4/Aliskiren/KTx
Record Dates: First submitted 2015-05-08; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Albuminuria
Keywords: direct renin inhibitor; kidney transplantation; albuminuria
MeSH Terms: conditions — Albuminuria | interventions — aliskiren; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- aliskiren - placebo - losartan (Experimental): aliskiren (Rasilez) 150 mg; losartan (Xartan) 50 mg
  Interventions: Drug: aliskiren; Drug: losartan; Other: Placebo
- losartan - placebo - aliskiren (Experimental): aliskiren (Rasilez) 150 mg; losartan (Xartan) 50 mg
  Interventions: Drug: aliskiren; Drug: losartan; Other: Placebo

INTERVENTIONS:
Drug: aliskiren — aliskiren will be administered at a dose of 150 mg, each dose was to be taken orally with water once daily at approximately 8:00 A.M., except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed. Drug compliance will be assessed by tablet counts.
  Other Names: Rasilez (Novarits Europe)
Drug: losartan — losartan will be administered at a dose of 50 mg, each dose was to be taken orally with water once daily at approximately 8:00 A.M. except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed. Drug compliance will be assessed by tablet counts.
  Other Names: Xartan (Adamed, Poland)
Other: Placebo — placebo will be administered once daily orally (1 tablet) in the morning with water at approximately 8:00 A.M. except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed. Compliance will be assessed by tablet counts. Placebo was prapared in Department of Pharmaceutical Technology MU Gdańsk

SUMMARY:
The study is a randomised, double-blind, controlled 2 x 3 cross-over trial in which the renal effects of therapy with aliskiren (A), placebo (P) and losartan (L) will be compared. It consists of an 8-week run-in period, 8 weeks of active treatment with aliskiren or losartan (period 1), 8 weeks of active treatment with the alternative medication (period 2), and an 8-week placebo administration between them.

DETAILED DESCRIPTION:
At the beginning, subjects who met the inclusion criteria will enter the 8-week run-in screening period. All hypotensive group of drugs will be allowed with exception of ACEI, ARA, DRI and mineralocorticoid receptor antagonists. The target BP will be an office trough BP of 140/90 mmHg or less. At the end of the run-in period, patients will be randomly allocated to one of the two treatment sequences: L/P/A (sequence 1) or A/P/L (sequence 2) . The study medications will be introduced as single hypotensive drug or added to the current hypotensive agents, the dosage of which, once adjusted in the run-in period, will be left unchanged throughout the study. Losartan will be used at a dose of 50 mg and aliskiren will be administered at a dose of 150 mg. Drug compliance will be assessed by tablet counts. Patients will be recommended not to change their usual daily protein and sodium intake during the study period. Dosage of cyclosporine or tacrolimus will be not allowed to change either. At the end of each of the three treatment periods, office thorough BP, 24-h ambulatory BP, albuminuria, serum creatinine and potassium, haemoglobin, cyclosporine or tacrolimus level, urine excretion of NAG, TGF-β-1 and 15-F2t-isoprostanes will be determined. eGFR will be calculated. Patients will be also asked to fill in the questionnaire for measuring patients-reported side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Transplantation period above 6 months,
2. Calcineurin inhibitor (cyclosporine or tacrolimus) based immunosuppression,
3. Stable cyclosporine or tacrolimus trough level in the last three months (no variations above 25%),
4. Stable renal function defined as eGFR > 30 ml/min (no variations above 5 ml/min/1.73 m2 in the last 3 months),
5. Arterial hypertension treated with one or two antihypertensive agents or blood pressure (BP) > 130/80 mmHg in patients not treated yet,
6. Albuminuria > 30 mg/g creatinine.

Exclusion Criteria:

1. Pregnant or the possibility of becoming so and breast feeding.
2. Angioedema from an ACE inhibitor or ARA in the history.
3. Serum potassium greater than 5.5 mmol/l on two or more occasions in the preceding three months.
4. Graft artery stenosis (i.e. psv of more than 200 cm/s in doppler usg)
5. Left ventricular dysfunction that requires an ACE inhibitor or an ARA Protocol Version 1 p. 5 of 10
6. New immunosuppressive agent was started or previous immunosuppressant stopped in the three months prior to study entry or plan to switch immunosuppressive agents within next three months.
7. Currently on four or more blood pressure pills and have an average blood pressure over three visits greater than 150/100.
8. Currently on an ACE-inhibitor or an ARAor treatment with an ACE inhibitor or ARA after kidney transplantation lasted more than 3 months.
9. Had an acute coronary syndrome, episode of malignant hypertension, stroke or transient ischaemic attack in the three months prior to study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
a difference in albuminuria in the measurements available for each patient | after 8 weeks of treatment

SECONDARY OUTCOMES:
a differences in N-acetyl-β-D-glucosaminidase (NAG) urine excretion in the measurements available for each patient | after 8 weeks of treatment
a differences in transforming growth factor β-1 (TGF-β-1) urine excretion in the measurements available for each patient | after 8 weeks of treatment
a differences in 15-F2t-isoprostanes (isoprostanes) urine excretion in the measurements available for each patient | after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boleslaw Rutkowski, Prof., Principal Investigator — Deaprtment of Nephrology, Transplantology and Internal Medicine, Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Gdansk, Pomeranian Voivodeship, Poland

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471